CLINICAL TRIAL: NCT06519396
Title: Ultrasonographic Achilles Tendon Measurements and Static and Dynamic Balance in Prediabetes
Brief Title: Achilles Tendon and Balance in Prediabetes
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Onur Armağan, Medical doctor, Prof., Eskisehir Osmangazi University
Other Study IDs: Achilles
Record Dates: First submitted 2024-05-31; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: PreDiabetes
Keywords: Achilles Tendon; Balance; Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients in the control group had FPG< 100 mg/dl or 75g oral glucose tolerance test: second hour plasma glucose <140mg/dl and HbA1c values <5.7%.
  Interventions: Device: ultrasonography evaluation; Device: tetrax device evaluation
- Prediabetes: The diagnosis of prediabetes was also confirmed through the patients' medical records. Patients with FPG 100-125 mg/dl or 75g oral glucose tolerance test: second hour plasma glucose 140-199 mg/dl and HbA1c values 5.7-6.4% was included in the prediabetes group.
  Interventions: Device: ultrasonography evaluation; Device: tetrax device evaluation
- Diabetes: The diagnosis of Type 2 Diabetes was confirmed through the patients' medical records. Patients with FPG≥ 126mg/dl or 75g oral glucose tolerance test: second hour plasma glucose ≥200mg/dl and HbA1c ≥6.5% were included in the diabetes group.
  Interventions: Device: ultrasonography evaluation; Device: tetrax device evaluation

INTERVENTIONS:
Device: ultrasonography evaluation — Ultrasonographic measurements of the Achilles tendon were taken using Samsung Sonoace X7 ultrasound system equipped with an 8-13MHz linear transducer. After assuming a prone position on the examination table, the patients placed their feet against the wall and flexed their ankles to ensure optimal contact between the probe and the tendon. Measurements were taken separately on the right and left sides for each patient. Initially, the probe was positioned perpendicular to the long axis of the tendon for an axial plane assessment, followed by measurements of thickness (anterior-posterior), width (medial-lateral), and area at the level of the medial malleolus. The thickness and width measurements utilized the tendon's major axes, while the area measurements were automatically calculated by the device through continuous tracing of the tendon circumference in the same section
Device: tetrax device evaluation — A Tetrax device was used to assess static balance. The patient was positioned on the platform and subjected to tests in eight different positions. For each position, a test measurement was made for a duration of 32 seconds, for a total of approximately 5 minutes. The normal eyes-open position was taken as the reference. The effects of vision on balance were observed in the eyes-closed position. Balance is dependent on the back of the heels and the lower vertebrae in this position. Conversely, in the eyes-closed position with the head tilted 30 degrees forward, there is a load on the upper vertebrae and neck. Following the measurements, the Tetrax software program was used to calculate the Fall Index and Stability Index

SUMMARY:
The aim was to evaluate the Achilles tendon size and static and dynamic balance, as well as the role of Achilles tendon on balance in prediabetes. A total of 96 patients were divided into three groups: 1)the control group, consisting of patients without diabetes; 2)the prediabetes group; 3)the diabetes mellitus group. Ultrasonographic measurements of Achilles tendon sizes were performed. Dynamic balance was assessed using the Berg Balance Scale, static balance was assessed.The Self-Leeds Assessment of Neuropathic Symptoms and Signs was utilized to identify neuropathic pain.

DETAILED DESCRIPTION:
Background/Aims: There is a lack of studies that examine balance problems and Achilles tendon thickness in prediabetes, despite their common occurrence in diabetes. The aim was to evaluate the Achilles tendon size and static and dynamic balance, as well as the role of Achilles tendon on balance in prediabetic patients.

Methods: A total of 96 patients were divided into three groups: 1)the control group, consisting of patients without diabetes; 2)the prediabetes group; 3)the diabetes mellitus group. Ultrasonographic measurements of Achilles tendon sizes (thickness, width and area) were performed. Dynamic balance was assessed using the Berg Balance Scale, static balance (the Fall Index, Stability Indexes) was assessed using a Tetrax device. The Self-Leeds Assessment of Neuropathic Symptoms and Signs was utilized to identify neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* being between 40 and 65 years old

Exclusion Criteria:

* extremity amputation
* vitamin B12 deficiency
* Type 1 Diabetes Mellitus
* prior exposure to neurotoxic agents
* peripheral neuropathy for reasons such as chronic kidney failure, liver failure, - hypothyroidism, hereditary and inflammatory peripheral neuropathies, neuromuscular diseases, malignancies
* anti-neuropathic drug usage
* radiculopathy
* nerve trauma or surgery
* vasculitis and autoimmune disorders
* peripheral vascular disease
* pregnancy
* vestibular and cerebellar problems
* history of lower extremity surgery
* presence of medication affecting balance
* history of alcoholism
* presence of visual impairment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study was conducted with 90 patients who were admitted to a Physical Medicine and Rehabilitation outpatient clinic. The patients were divided into three groups: 1) the control group (patients who were neither prediabetic nor diabetic; 2) the prediabetes group (prediabetic patients); and 3) the Diabetes Mellitus group (patients with Type 2 Diabetes Mellitus).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement of achilles tendon | baseline
  measurements of thickness (anterior-posterior), width (medial-lateral), and area of achilles tendon at the level of the medial malleolus were made
balance measurement | baseline
  Static balance measurement were made with Tetrax Device

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakilan, Study Director — Eskişehir Osmangazi University
Locations (1):
- Fulya Bakilan, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No